CLINICAL TRIAL: NCT04546711
Title: Effects of Ketogenic Diet on Epilepsy: Metabolism and Quality of Life
Brief Title: Energy Expenditure and Quality of Life in Epilepsy
Status: Withdrawn | Type: Observational
Why Stopped: decided not to process with study
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-0371; A535100 (Other: UW Madison); SMPH/NEUROLOGY/NEUROLOGY (Other: UW Madison); Protocol Version 4/27/2020 (Other: UW Madison)
Record Dates: First submitted 2020-09-04; First posted 2020-09-14 (Actual); Last update posted 2023-06-29 (Actual); Status verified 2023-06

CONDITIONS: Epilepsy
Keywords: Ketogenic Diet; Quality of Life; Energy Metabolism; Physical Activity
MeSH Terms: conditions — Epilepsy; Motor Activity | interventions — Diet, Ketogenic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Ketogenic Diet: * Baseline Assessments
  * Ketogenic diet intervention
  * 3 and 6 month Assessments
  Interventions: Other: Ketogenic Diet

INTERVENTIONS:
Other: Ketogenic Diet — The ketogenic diet (KD) is a high fat, very low carbohydrate diet

SUMMARY:
The main objectives of this study are to investigate the influence of the ketogenic diet (KD), standard care for patients assisted in the UW Health Adult Epilepsy Dietary Therapy Clinic, on changes in the frequency and severity of seizures, QoL, energy substrate metabolism, body energy expenditure components, fat mass and fat-free mass in adults with epilepsy. To achieve this objective, twenty-five male and female participants between the ages of 18 and 45 years (or over 18 years for remote participation), who accepted to initiate the KD as a standard of care prescribed by their physician, will be recruited according to inclusion/exclusion criteria. Participants will be on study for 6 months.

DETAILED DESCRIPTION:
The ketogenic diet (KD) is a high fat, very low carbohydrate diet that promotes a variety of changes in the chemical processes on the body associated with reduced frequency and severity of seizures in patients with epilepsy. The reasons for this improvement are not yet fully understood and the answers can be related to changes in the biochemical process and the use of different substrates as the main source of energy for the body.

The quality of life (QoL) of patients with epilepsy is highly affected by stigmatization, difficulties with employment, and physical limitations. There is some evidence that the KD may have beneficial effects on QoL in patients with epilepsy, which can be investigated by changes in body energy expenditure (e.g. physical activity level). Studies that associate changes in body energy requirements, body composition and biochemical measures with seizures and QoL are currently limited in the scientific literature.

The main objectives of this study are to investigate the influence of the KD on changes in the frequency and severity of seizures, QoL, energy substrate metabolism, body energy expenditure components, fat mass and fat-free mass in adults with epilepsy. To achieve this objective, twenty-five male and female participants between the ages of 18 and 45 years (or over 18 years old for remote participation, no metabolic analysis will be complete on remote participants) will be recruited according to inclusion/exclusion criteria. Data will be collected at baseline (time of enrollment), and again at 3 and 6 months following diet start. Stable isotope compounds (doubly labeled water) will assess total daily energy expenditure (TDEE) and body composition (fat mass; fat-free mass). Indirect calorimetry will assess the resting energy expenditure (REE) and respiratory quotient for energy substrate oxidation. Biochemical blood exams (fasting glucose and insulin, and ketone bodies) and anthropometric data will provide data on the nutritional and metabolic status of the participant. Seizure frequency, severity, and QoL will be evaluated using validated self-report questionnaires. The physical activity level, obtained through the ratio between TDEE and REE and by wearing of a physical activity monitor, will be used as a predictor of QoL.

The hypothesis is that KD therapy promotes differences in energy metabolism and energy substrate oxidation, which will lead to better metabolic control of epilepsy, reduced frequency and severity of seizures, and also an improved patient QoL. This study is expected to help elucidate the metabolic changes associated with reduced seizure frequency and severity, and improvement of QoL in patients with epilepsy.

ELIGIBILITY:
Inclusion Criteria (in person participation):

* aged 18-45
* Diagnosis of epilepsy
* Experience an average of 2 or more seizures per month during the 3 months prior to study
* Plan to start oral ketogenic diet therapy (e.g. with the modified Atkins diet)
* Have low average or higher cognitive/intellectual function and are able to complete self-report questionnaires

Inclusion Criteria for Remote Participation:

* over 18 years of age (no age limit)
* Diagnosis of epilepsy
* Experience an average of 2 or more seizures per month during the 3 months prior to study
* Plan to start oral ketogenic diet therapy (e.g. with the modified Atkins diet)
* Have low average or higher cognitive/intellectual function and are able to complete self-report questionnaires

Exclusion Criteria:

* Participants who report being claustrophobic
* Presence of edema, conditions or persistent side effects of medication use (e.g. vomiting, diarrhea, excessive sweating, and burns) that could cause alterations in the body hydration and consequently, be a bias in energy metabolism variables
* Currently using medications that may cause metabolic and/or absorptive alterations (e.g. diuretics, amphetamines, lipase inhibitors, corticosteroids, etc.)
* Unstable metabolic condition (e.g. persistent sodium <130 or glucose <50)
* Liver, kidney, or pancreatic disease
* Hypercholesterolemia (cholesterol > 300mg/dL)
* Currently pregnant or planning on becoming pregnant
* Fatty acid oxidation disorder or pyruvate carboxylase deficiency
* Already on ketogenic therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 25 male and female adults between the ages of 18-45 (for in person participation) and over 18 (for remote participation) with epilepsy.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2023-06 (Estimated); Primary Completion 2025-08 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Change in the Frequency of Seizures Assessed with Participant Seizure Frequency Report | baseline, 3 months, 6 months
  The hypothesis is that participants will have a significant reduction in seizures (>50%) at 3 and 6 months following the start of KD therapy.
Change in Severity of Seizures Assessed by Seizure Severity Questionnaire (SSQ) | baseline, 3 months, 6 months
  The SSQ scores range from 1-7 with lower scores indicating improved status. The hypothesize is that participants will have a significant reduction in seizures (>50%) at 3 and 6 months following the start of KD therapy, which will also lead a significant reduction (p<0.05) of SSQ overall score.
Change in the Quality of Life in Epilepsy (QOLIE-31-P) Score | baseline, 3 months, 6 months
  The QOLIE-31-P instruments include seven multi-item scales that tap the following health concepts: emotional well-being, social functioning, energy/fatigue, cognitive functioning, seizure worry, medication effects, and overall quality of life. The total range of possible scores is 0-100, higher scores indicate better well being. The hypothesis is that participants will have a significant reduction in seizures (>50%) at 3 and 6 months following the start of KD therapy, which will also lead to significant improvement (p<0.05) in the QoL overall score.

SECONDARY OUTCOMES:
Enhanced Metabolic Control of Epilepsy Assessed by Indirect Calorimetry | baseline, 3 months, 6 months
  The hypothesis is that KD therapy will promote significant differences (compared to pre-diet baseline) in substrate oxidation (an increase in fat oxidation and a decrease in carbohydrate oxidation) which will correlate with seizure reduction.
Change in Physical Activity Level (PAL) as Recorded by Actigraph Measurement | baseline, 3 months, 6 months
  The hypothesis is that KD therapy will contribute to an increase of PAL (direct contribution of KD), leading to an increase of total daily energy expenditure (TDEE) (indirect contribution of KD).
Change in Body Fat Mass | baseline, 3 months, 6 months
  The hypothesis is that KD therapy will contribute to a decrease in fat mass, a maintenance of fat-free mass.

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Felton, MD, PhD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No